CLINICAL TRIAL: NCT06735950
Title: The Volunteering-in-Place Program for Apathetic Assisted Living Residents With ADRD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jennifer Klinedinst, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HP-00112822; 1R61AG088468-01A1 (NIH)
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Apathy in Dementia
Keywords: apathy; assisted living; dementia; volunteering
MeSH Terms: conditions — Lethargy; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Volunteering-in-Place Program (Experimental): Participants in this arm will engage in a volunteer activity in the assisted living facility chosen based on their interests and capabilities.
  Interventions: Behavioral: Volunteering in Place Program
- Recreational Activity (Active Comparator): Participants in this arm will engage in a current events group
  Interventions: Behavioral: Recreational activity

INTERVENTIONS:
Behavioral: Volunteering in Place Program — Implementation of the VIP Program consists of 4 steps guided by the Social Ecological Model (SEM) with Interpersonal interventions guided by Social Cognitive Theory (SCT), and will be implemented over a 6-month period by research supported Volunteer Coordinators. The four steps of the VIP Program are: Step 1: Stakeholder Team, Staff and Family Education; Step 2: Assessment of AL Environment and Residents Abilities and Interests; Step 3: Ongoing Implementation of the Volunteer Plan; and Step 4: Reassessment of the Volunteer Activity. Participants will volunteer three time per week for approximately 30 minutes.
  Other Names: VIP Program
  Arms: Volunteering-in-Place Program
Behavioral: Recreational activity — The Recreational Activities group intervention will consist of similar staff education regarding the benefits of engaging residents in meaningful activities as described in Step 1 above, without other steps associated with the VIP Program. The Recreational Activities group will be exposed to a research team RA coordinator who will provide a current events activity (reviewing the daily newspaper) for the participants in the RA group three times per week for approximately 30 minutes as an attention control.
  Other Names: Current events group
  Arms: Recreational Activity

SUMMARY:
This is a research study to test two different interventions to decrease apathy in assisted living residents with some memory issues. Apathy makes older adults not feel like doing much activity. This study is completely voluntary and will not affect the care you receive at your assisted living community.

The two possible interventions are 1) participation in a volunteering opportunity within the assisted living community OR 2) participation in a guided current events group within the assisted living community. These activities would be in addition to any other regular activities you participate in within the assisted living community. Both activities would take place three days per week for approximately 30 minutes. You would be randomly assigned (like a coin flip) to which intervention you would do. You do not get to choose. You would participate in the activity for a total of 6 months.

In addition to participating in the intervention (either volunteering or current events), you will be asked to answer some questions about your memory, level of activity, mood, confidence in your ability to do a volunteer job, and feelings of usefulness. You will answer these questions at baseline (before the activity begins, at 3 months after doing the intervention activity, and aging at 6 months after starting the interventions activity. You will also be asked to wear a MotionWatch for 5 days at each time point (baseline, 3months and 6 months). A motion watch measures your level of activity. It feels like wearing a regular watch. You will be in the study for 6 months total.

Risks to participating in this study are minimal and include privacy (other people may find out you are in the study), confidentiality of the data collected if someone other than study staff accesses your records, fatigue with answering the questionnaires, and some mild discomfort with wearing the MotionWatch. This is also a minor risk that you could fall or otherwise harm yourself getting to or participating in your intervention activity.

The benefit of participating in this study include possible enjoyment of participating in the intervention activity.

DETAILED DESCRIPTION:
Our Primary aim is to test the preliminary efficacy of the VIP Program to decrease apathy and sedentary activity among apathetic AL residents with mild to moderate ADRD at 3 and 6 months post implementation. Hypothesis 1.1: Participants in the VIP Program will have a decrease in apathy and a decrease in time spent in sedentary activity when compared to residents exposed to RA only at 3 and 6 months post implementation of the intervention. This study will use a cluster randomized control trial with a repeated measures design. A total of 4 AL communities will be randomized to treatment [Volunteering-in-Place (VIP) Program intervention] or time equivalent control [current events group]. Randomization will occur via random number generator at the facility level rather than at the individual level in order to control for carryover of VIP Program activities. Data will be collected at baseline, 3 and 6 months post initiation of the VIP Program. The 3 month time point was chosen as it takes at least three months for the VIP Program interventions to become ingrained into the residents routine and to impact apathy outcomes. We will assess for effects at 6 months as this time point is indicative of longer-term behavior change and evidence of sustainability of the program and resident and staff participation.

The Assisted Living communities included in this study will be located in the State of Maryland. We will randomly select from the 10 total AL communities across these provider organizations to contact and enroll specific sites. To be eligible to volunteer to participate in the study the AL community will need to: (1) have at least 100 beds; and (2) identify a stakeholder team and champion to work with us throughout the study period. AL communities will be excluded if they have an existing in-house volunteer program for residents with ADRD.

Potential participants will have an opportunity to learn about the study via the resident and family information sessions.

Resident recruitment will be done in person by obtaining a list of all potentially eligible residents from a designated staff member and randomly approaching each resident until 27-28 residents per setting are fully enrolled by research team evaluators. Residents who meet initial inclusion criteria will be given an Evaluation to Sign Consent and if they pass they will continue with the full consent process. If they do not pass the Evaluation to Sign Consent, they will be asked to verbally provide assent and the Legally Authorized Representative will be approached to complete the consenting process.

Once consent is obtained, cognitive testing and an apathy screening will be done by a trained evaluator to determine eligibility. Residents will be considered to have mild to moderate ADRD if they have a score of 26 or below on the Saint Louis University Mental Status Exam (SLUMS) and can follow a one step command ("touch your nose"). The evaluator will collect the data on the SLUMS and assess the ability to follow a one step command from the resident. Once eligibility for cognitive impairment has been established, a family member or a direct care worker familiar with the participant's behavior over the past month would complete the Neuropsychiatric Inventory (NPI) apathy subscale about the resident. Residents who have a "yes" answer to at least 2 questions on the apathy subscale of the NPI will be enrolled.

Implementation of the VIP Program consists of 4 steps guided by the Social Ecological Model (SEM) with Interpersonal interventions guided by Social Cognitive Theory (SCT), and will be implemented over a 6-month period by research supported Volunteer Coordinators. Each part of the SEM addresses a portion of the resident, caregiver and environmental stressors that contribute to apathy. The Volunteer Coordinators will have experience working with older adults with ADRD. The Volunteer Coordinator will work 20 hours per week for the 6-month intervention period. In addition, the Volunteer Coordinator will work with the stakeholder team to identify a Staff Champion to work with the Volunteer Coordinator on the VIP Program to optimize implementation and assure sustainability. The Volunteer Coordinator and Staff Champion will meet monthly with the stakeholder team to make sure that the resident volunteer activities are supported by the facility employees and to problem solve any challenges related to the VIP Program (e.g., resistance of staff to help residents get to volunteer activities).

Separate interventionists will be used for the Recreational Activities Only (current events) group to prevent crossover effects. The Recreational Activities group intervention will consist of similar staff education regarding the benefits of engaging residents in meaningful activities as the VIP intervention, without other steps associated with the VIP Program. Prior research has repeatedly demonstrated that education alone in these settings is insufficient to alter staff or resident behavior. The Recreational Activities group will be exposed to a research team RA coordinator who will provide a current events activity (reviewing the daily newspaper) for the participants in the RA group three times per week for approximately 30 minutes as an attention control. This control intervention provides some opportunity for engagement in activities but there is no development of a person-centered volunteer activity that is meaningful to the individual and no interventions to strengthen self-efficacy expectations about volunteering or participating and no focus on imparting feelings of usefulness as the mechanism to decrease apathy. Moreover, it is consistent with usual types of activities provided in AL.

Data will be collected at baseline, 3 and 6 months. All data will be collected by a trained research evaluator.

AL Facility Descriptive Data: AL facility size, staffing levels (number of RNs, LPNs, direct care workers, activity staff), and highest level of care provided (level 1, 2, 3) will be obtained at baseline from the AL Administrator or designee for each community and will be considered as covariates.

Once enrolled: Resident participants will complete baseline questionnaires with input from a direct care worker if necessary. These questionnaires include the Apathy Evaluation Scale, the Yale Physical Activity Survey-Recreational activity subscale modified for assisted living residents, the Cornell Scale for Depression in Dementia, three questions on feelings of usefulness, and three questions on self-efficacy or volunteering. In addition, participants will wear a motion watch (accelerometer) for 5 weekdays to assess sedentary behavior. These questionnaires and Motion watch measures will be repeated at 3 post intervention and 6 months post intervention. At baseline, we will collect descriptive data including resident age, race, gender, ethnicity, marital status, length of time residing in AL, and education from the AL clinical record. At each time point, we will also collect medications, comorbidities - using the Cumulative Illness Rating Scale, falls, hospitalizations, emergency room visits and transfers to a higher level of care such as a skilled nursing facility.

Participants randomized to the VIP Program:

After completing baseline measures, residents in the VIP Program intervention will meet with the Volunteer Coordinator (interventionist) and/or Staff Champion (AL staff member interventionist) at a mutually convenient day/time for an assessment of their Interests, Physical Capability Scale and for input regarding their volunteer plan. (VIP Program Step 2) This should take approximately 30 minutes, but could be divided into multiple sessions to provide breaks for the resident. Once the resident and Volunteer Coordinator decide on a volunteer activity and plan, the resident will begin volunteering 3 days per week for 30 minutes each time for 6 months. (VIP Program Step 3) The Volunteer Coordinator and other staff will implement the appropriate self-efficacy based motivational strategies. The Volunteer Coordinator and/or Staff Champion will elicit feedback from the resident regarding their enjoyment of the volunteer activity using the Resident Evaluation of Volunteer Experience form. However, residents will be encouraged to provide feedback regarding the activity to the Volunteer Coordinator any time they desire or are not happy with the activity for any reason. The Volunteer Coordinator or Staff Champion will make adjustments to the Volunteer Activity or address any issues with input from the resident, study staff and stakeholder team.

For Participants in the Recreational Activities Control Group:

The Recreational Activities group intervention will consist of similar staff education regarding the benefits of engaging residents in meaningful activities as described in Step 1 above, without other steps associated with the VIP Program. Separate interventionists will be used for the VIP vs. Recreational Activities groups to reduce crossover effects. Prior research has repeatedly demonstrated that education alone in these settings is insufficient to alter staff or resident behavior. The Recreational Activities group will be exposed to a research interventionist who will provide a current events activity (reviewing the daily newspaper) for the participants in the RA group three times per week for approximately 30 minutes as an attention control. This control intervention provides some opportunity for engagement in activities but there is no development of a person-centered volunteer activity that is meaningful to the individual and no interventions to strengthen self-efficacy expectations about volunteering or participating and no focus on imparting feelings of usefulness as the mechanism to decrease apathy. Participation in the current events activity will be tracked for treatment fidelity using the same Participation Index as the VIP Program intervention.

ELIGIBILITY:
Inclusion Criteria:

* age 55 years or older;
* English speaking;
* live in the included AL community
* have mild to moderate cognitive impairment based on a SLUMS score of 26 or below and the ability to follow a one-step command.
* have apathy based on a "yes" answer to at least 2 questions on the apathy subscale of the Neuropsychiatric Inventory (NPI) completed by a family or staff member who has had close contact with the resident in the past month;
* have an anticipated length of stay of 12 months.

Exclusion Criteria:

- refusal to assent

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Apathy Evaluation Scale | Baseline, 3 months, 6 months
  The Apathy Evaluation Scale-Informant (AES-I) will be used to assess apathy. The AES-I has 18 items that assess cognitive, behavioral, and emotional aspects of apathy. The scale has good psychometric properties when used to assess apathy in adults with dementia. The total score ranges from 18 to 72, with higher scores indicating more apathy.

SECONDARY OUTCOMES:
Motion Watch | Baseline, 3 months, 6 months
  Objective sedentary activity will be obtained using three full weekdays of data from the MotionWatch 8©, a lightweight waterproof wrist worn tri-axial accelerometer that reliably measures activity in 60 second epochs of time.98 The resident will wear the MotionWatch for five days and the first and last day of data will not be included so as to get three complete days of data. The MotionWatch 8© contains a miniature accelerometer to allow measurement and recording of physical movement of the wrist which provides a close correlation to whole body movement. Reliability, validity, and cut points for different levels of activity have been established for older adults. Specifically we will collect counts of activity and time spent in sedentary activity during weekdays where the volunteer activity or recreational activity took place as this is when we expect to see changes in sedentary activity.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Klinedinst, PhD, MPH, RN, Principal Investigator — University of Maryland, Baltimore

IPD SHARING:
Plan to Share IPD: Yes
Data will be deposited in a data repository after the completion of the study.
Time Frame: after the conclusion of the study data will be stored in the repository indefinitely
Access Criteria: People with access to the specified repository.